CLINICAL TRIAL: NCT01244113
Title: Optimal Dose of Propofol for Induction of Deep Sedation for Brain MRI Scanning in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Hae-Keum Kil / Proffesor, Severance Hospital, Department of Anaesthesiology and Pain Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 4-2010-0150
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: propofol — optimization of propofol dose from 1.5 mg/kg to 2.5 mg/kg using Dixon's up and down method during MRI scanning

SUMMARY:
The children with CP has been shown different drug responses from the normal population of children and it may related with a various oral medications such as baclofen, tizanidine, diazepam, dantrolene, or anticonvulsant drugs.

The aim of this study is to establish the optimal induction dose of propofol for deep sedation to start MRI for < 30 min in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* children with cerebral palsy with patient agreement

Exclusion Criteria:

* sleep apnea, difficult airway, cardiorespiratory disease, allergic history to propofol

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Keum Kil, MD, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea